CLINICAL TRIAL: NCT04634578
Title: Bevacizumab Treatment For Type 1 Retinopathy of Prematurity
Brief Title: Bevacizumab Treatment For Type 1 ROP
Acronym: ROP4
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ROP4; UG1EY011751 (NIH)
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bevacizumab- 0.063 mg (Experimental): Participants will receive a single intravitreal injection of 0.063 mg of bevacizumab in one or both eyes following enrollment into the study. The injection/s should be given as soon as possible but no later than 2 days after the diagnosis of type 1 ROP meeting all of the inclusion criteria and none of the exclusion criteria.
  Interventions: Drug: Bevacizumab
- Bevacizumab- 0.25 mg (Experimental): Participants will receive a single intravitreal injection of 0.25 mg of bevacizumab in one or both eyes following enrollment into the study. The injection/s should be given as soon as possible but no later than 2 days after the diagnosis of type 1 ROP meeting all of the inclusion criteria and none of the exclusion criteria.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — All participants will receive a single intravitreal injection of bevacizumab in one or both eyes following enrollment into the study. The injection/s should be given as soon as possible but no later than 2 days after the diagnosis of type 1 ROP meeting all of the inclusion criteria and none of the exclusion criteria.
  Eyes meeting eligibility criteria will receive a single dose of 0.063 mg or 0.25mg bevacizumab provided by the pharmacy at the investigator's institution.
  Other Names: Avastin

SUMMARY:
Type 1 retinopathy of prematurity in zone I represents the most severe type of ROP and has the worst prognosis. It is unknown whether low-dose bevacizumab will be successful in these severe cases. Also unknown is the timing and extent of peripheral retinal vascularization after low-dose bevacizumab compared with the standard dose. The current study will evaluate whether doses of 0.063 mg and 0.25mg are effective as treatment for type 1 ROP, with ROP and retinal vessels all in zone I.

DETAILED DESCRIPTION:
Infants with type 1 ROP and no prior treatment for ROP will be randomly assigned (1:1) to treatment with either intravitreous bevacizumab 0.063 mg or either intravitreous bevacizumab 0.25 mg. Study exams will be at 1 day, 4 days (if no improvement on day 1), 1, 2, 3, and 4 weeks, and at 2 and 4-months post-treatment (and re-treatment when indicated). Additional study exams will occur at adjusted age 6 and 12 months. Non-study examinations will be at clinician discretion and are likely to occur more often. The primary outcome will be treatment success within each dose group, defined as improvement by the day 4 exam and no recurrence of type 1 ROP or severe neovascularization requiring additional treatment within 4 weeks of injection. Important secondary outcomes include safety and efficacy. refractive outcomes, and the extent of retinal vascularization at 2 and 4 months post-injection between the two dose groups.

ELIGIBILITY:
Inclusion Criteria:

The study participant must have at least one eye meeting all of the inclusion criteria in order to be eligible to participate:

1. Birth weight < 1251 grams
2. Newly diagnosed (within 2 days) type 1 ROP in zone I in one or both eyes

Exclusion Criteria:

Participants meeting any of the following exclusion criteria will be excluded from study participation.

1. Previous treatment for ROP
2. Stage 4 or 5 ROP in either eye
3. Treatment could not be done within 2 days of diagnosis of type 1 ROP
4. Investigator unwilling to randomize or parent unwilling to accept randomized assignment to either treatment
5. Transfer to another hospital anticipated within the next 4 weeks where exams by study-certified examiners are not available. If hospital discharge is anticipated within the next 4 weeks, parents unable or unwilling to return to the PEDIG site for outpatient follow-up visits.
6. Active ocular infection or purulent nasolacrimal duct obstruction in either eye

One eye will be excluded, and other eye may be eligible, if either of the following are present:

* Visually significant ocular anomaly (e.g., cataract, coloboma)
* Opacity that precludes an adequate view of the retina

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Success at 4 Weeks Post Injection | 4 weeks
  Treatment success, determined at 4 weeks, post injection, and meeting all the following criteria:
  * Improvement by the 4-day exam (3 to 5 days)
  * No recurrence of type 1 ROP or severe neovascularization requiring additional treatment within 4 weeks of injection.

CONTACTS AND LOCATIONS:
Overall Officials: David K Wallace, MD, MPH, Study Chair — Vanderbilt University
Locations (26):
- United States (25):
  - Arkansas Childrens Hospital/ University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Univ of California, Irvine- Gavin Herbert Eye Institute, Irvine, California
  - Jules Stein Eye Institute at the University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California San Francisco Department of Ophthalmology, San Francisco, California
  - The Emory Eye Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - U of Illinois at Chicago Eye and Ear Infirmary, Chicago, Illinois
  - University of Chicago, Hyde Park, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - UK Ophthalmology and Visual Sciences, The Eye Clinic, Lexington, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - New York Presbyterian David H Koch Center, New York, New York
  - Duke University Eye Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Pediatric Ophthalmology Associates, Inc., Columbus, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Eye Center of Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Storm Eye Institute, Mt. Pleasant, South Carolina
  - Texas Children's Hospital - Dept. Of Ophthalmology, Houston, Texas
  - University of Utah Moran Eye Center, Salt Lake City, Utah
  - Virginia Pediatric Eye Center, Norfolk, Virginia
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the Pediatric Eye Disease Investigator Group (PEDIG) public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after publication of each primary manuscript.
Access Criteria: Users accessing the data must enter an email address.

REFERENCES:
- See also: PEDIG Public Website — https://public.jaeb.org/pedig

DOCUMENTS (3):
  • Study Protocol (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT04634578/Prot_007.pdf
  • Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT04634578/SAP_001.pdf
  • Informed Consent Form (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT04634578/ICF_006.pdf